CLINICAL TRIAL: NCT02969902
Title: Randomized Controlled Trial to Compare Buzzy and Hand-held Computer Distraction for Pain Control in Children Underwent Venipuncture.
Brief Title: Buzzy Distraction During Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Luca Ronfani, Head of Clinical Epidemiology and Public Health Research Unit, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 19/13
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Pain Relief
Keywords: Procedural pain; Phlebotomy; Distraction; Hand-held computer; Children
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy® device (Experimental): The Buzzy® device is applied just above the selected site of the venipuncture; an ice pack is attached under the device; the device is turned on and after 15 second the venipuncture is made.
  Interventions: Device: Buzzy® device
- Hand-held computer (Active Comparator): Using an hand-held computer, children start to play with an age-appropriate videogame three minutes before the procedure. They continue to play during the venipuncture.
  Interventions: Device: Hand-held computer

INTERVENTIONS:
Device: Buzzy® device
  Arms: Buzzy® device
Device: Hand-held computer
  Arms: Hand-held computer

SUMMARY:
Venipuncture is one of the most common iatrogenic painful and stressful procedures performed on children. Interventions aimed at reducing the distress related to this experience are widely and strongly recommended. Pain and anxiety management is even more essential because it may modify children's memory for procedural pain and the subsequent acceptance of later health care painful interventions. Distraction is the most studied psychological technique to relieve venipuncture related pain and distress, with a strong evidence supporting its efficacy in children and adolescents.

In recent years several studies showed the effectiveness of a specific tool named Buzzy® (MMJ Labs, Atlanta GA, USA), in relieving pain and distress in children. Buzzy combines distraction and physical analgesia (vibration and cold) and it was positively tested during venipuncture, intravenous cannulation and painful injections in children. Even though its efficacy it's well established, most of the published trials did not compare Buzzy with other interventions, so that little data are available about its usefulness compared with other distractions techniques.

Hand-held computers are reusable tools, which offer a technological-based active distraction. There is evidence supporting their used during painful procedures such as venipuncture and a recent published study showed that hand-held computer distraction was as effective as nurse-led passive distraction techniques in children.

The aim of this study is to compare the effectiveness of Buzzy versus hand-held computer in pain relief during venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* children from 4 to 12 years of age needing venipuncture

Exclusion Criteria:

* the presence of damage, denuded or broken skin in the site of Buzzy application;
* use of topical, enteral or parenteral analgesics within eight hours before enrolment;
* the presence of cognitive impairment or the inability to report pain verbally;
* the presence of chronic disease, included epilepsy, or of diseases associated with cold hypersensitivity (i.e., sickle cell anaemia, Raynaud's disease).

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | Within 5 minutes after the procedure
  Children from 4 to 7 years of age record their pain using the Faces Pain Scale-Revised (FPS-R); children from 8 to 12 years using a Numerical Rating Scale, with scores from zero to 10.

SECONDARY OUTCOMES:
Pain evaluated by parents | Within 5 minutes after the procedure
  Pain evaluated using a Numerical Rating Scale, with scores from zero to 10
Pain evaluated by nurses | Within 5 minutes after the procedure
  Pain evaluated using a Numerical Rating Scale, with scores from zero to 10
Success at first attempt | Intraprocedural
  Percentage of success at first attempt
Adverse events | Up to 15 minutes after the procedure
  The number and the type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Chair — IRCCS Burlo Garofolo; Franca Crevatin, RN, Study Director — IRCCS Burlo Garofolo